CLINICAL TRIAL: NCT05854173
Title: Compare The Effect of Pendulum Exercises With the Kaltenborn Mobilization Among the Patients of Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/536
Record Dates: First submitted 2023-03-18; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pendulum Exercises (Other)
  Interventions: Diagnostic Test: Pendulum Exercises
- Kaltenborn Mobilization (Experimental)
  Interventions: Diagnostic Test: Kaltenborn Mobilization

INTERVENTIONS:
Diagnostic Test: Pendulum Exercises — Compare The Effect of Pendulum Exercises Among the Patients of Adhesive Capsulitis
  Arms: Pendulum Exercises
Diagnostic Test: Kaltenborn Mobilization — Compare The Effect of Kaltenborn Mobilization Among the Patients of Adhesive Capsulitis
  Arms: Kaltenborn Mobilization

SUMMARY:
To determine the effect of pendulum exercises with the kaltenborn mobilization among the patients of adhesive capsulitis

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be of the age group of 40-60 years.
* Can be male or female
* Diagnosed with adhesive capsulitis by orthopedic or physical therapist.
* Pain, stiffness, and limitation of passive shoulder lateral rotation, abduction, and internal rotation of more than 50% compared with the opposite side for at least 3 months

Exclusion Criteria:

* Presence of neurological disorders (e.g., stroke, Parkinson's disease) leading to deficiency of shoulder muscles activity, Severe trauma related to painful stiff shoulder which leads to bony changes of the affected shoulder on radiographs, Previous surgeries and manipulation under anesthesia of the affected shoulder

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain assessed by Visual Analog Scale | 6 Months
disability index | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University CRC, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No